CLINICAL TRIAL: NCT03374462
Title: Use of Home-Based Telemedicine to Improve Healthcare Utilization and Outcomes in Pediatric Patients With Poorly Controlled Type 1 Diabetes
Brief Title: Type 1 Diabetes Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1125857
Record Dates: First submitted 2017-11-27; First posted 2017-12-15 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine Intervention (Experimental): All participants will receive the study intervention, which consists of home-based telemedicine visits with a diabetes specialist, at a frequency determined by the patient's degree of glycemic control (every 4, 6, or 8 weeks).
  Interventions: Behavioral: Telemedicine Intervention

INTERVENTIONS:
Behavioral: Telemedicine Intervention — Home-based telemedicine visits

SUMMARY:
At the conclusion of this project, investigators will have assessed the effectiveness of home-based telemedicine for improving multiple important clinical and patient-centered outcomes in a high-risk pediatric cohort with T1D.

Aim 1. To test the hypothesis that home-based telemedicine is a feasible and acceptable method of care delivery for patients with poorly controlled type 1 diabetes (T1D) currently cared for at the University of California, Davis (UCD) Pediatric Endocrinology clinic. Specifically:

A) Patients and families choose to participate in telemedicine visits as a supplement to in-person care; B) Patients and families can utilize secure, internet-based platforms to upload and share glucose meter data and to establish an audio-video connection with a diabetes specialist in their home settings; C) Patients and families are satisfied with the experience of home-based telemedicine and would choose to receive future diabetes care via this modality.

Aim 2. To test the hypothesis that using home-based telemedicine, these patients can complete more frequent visits with a diabetes specialist than they previously completed via office visits alone.

Aim 3. To test the hypothesis that increased contact with a diabetes specialist via home-based telemedicine will lead to significant improvement in glycemic control for these patients.

Aim 4. To evaluate the effects of increased contact with a diabetes specialist via home-based telemedicine on high-cost health care utilization - specifically emergency department (ED) visits and diabetes-related hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* age 1-17 years
* known diagnosis of T1D
* >1 prior visit to the UC Davis Pediatric Endocrinology clinic (to avoid enrolling newly diagnosed patients)
* suboptimal glycemic control, defined as most recent hemoglobin A1C level of >8%
* access to the internet via a device with video and audio capability (e.g. computer, tablet, mobile phone)
* ability to connect their home glucose meter to an internet-capable device via Bluetooth or physical cable for the purpose of data uploading.

Exclusion Criteria:

* Patients and parents whose primary language is not English
* Patients who have Western Health Advantage health insurance

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Improvement in A1C Levels | 12-months
  Investigators will compare the mean pre-study and mean post-study A1C levels

SECONDARY OUTCOMES:
Increased visit frequency | 24-months
  Investigators will evaluate if offering telemedicine visits leads to increased visit frequency for these patients during the 12-month study period, when compared to the previous 12-months
Impact on high-cost health care utilization | 24-months
  Investigators will compare the mean number of ED visits and mean number of diabetes-related hospitalizations for patients in the cohort
Feasibility of home-based telemedicine | 12-months
  Investigators will evaluate the feasibility of home-based telemedicine for the patient population by the percent of eligible patients who enroll in the study and the percent of enrolled patients who complete the study
Acceptability of home-based telemedicine | 12-months
  Investigators will evaluate the acceptability of home-based telemedicine for the patient population by the percent of those completing the study who express satisfaction with the telemedicine experience.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Crossen, MD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No